CLINICAL TRIAL: NCT01979029
Title: Affection on Anastomotic Blood Flow and the Lymph Nodes Dissection Between Division at the Root of the Inferior Mesenteric Artery and Preserving the Left Colic Artery in Rectum Cancer Surgery
Brief Title: Study of the Preservation of the Left Colic Artery on Rectum Cancer Surgery
Acronym: POTLCAORCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jian Suo (Other)
Responsible Party: Sponsor-Investigator, Jian Suo, Headmaster, Dept.of General Surgery, The First Hospital of Jilin University
Organization: The First Hospital of Jilin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Left Colic Artery
Record Dates: First submitted 2013-10-25; First posted 2013-11-08 (Estimated); Results first posted 2016-06-06 (Estimated); Last update posted 2016-06-06 (Estimated); Status verified 2016-04

CONDITIONS: Rectum Cancer
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- preserving the left colic artery (Experimental): We preserve the left colic artery and resect the No. 253 lymph node during the rectal surgery.
  Interventions: Procedure: preserving the left colic artery
- not preserving the left colic artery (Experimental): We preserve the high ligation of the inferior mesenteric artery during the rectal surgery.
  Interventions: Procedure: not preserving the left colic artery

INTERVENTIONS:
Procedure: preserving the left colic artery — The root of the inferior mesenteric artery(IMA) was carefully dissected and the artery wall was exposed all the way to the bifurcation of the left colic artery(LCA) and the superior rectal artery (SRA), exposing the LCA from its root until the inferior mesenteric vein (IMV) was recognized. Subsequently, dissection was continued along the IMV up to the level of the root of the IMA. Then the sigmoid mesentery was transected from the root of the IMA to the IMV, and the IMV and the root of the SRA were ligated. Finally, the adipose tissue with the lymph nodes in the area surrounded by the IMA, IMV, and LCA was dissected, with preservation of the LCA .
  Arms: preserving the left colic artery
Procedure: not preserving the left colic artery — The root of the IMA was exposed and the fatty tissue around the root of the IMA was swept in order to maximize the lymph node retrieval rate. Subsequently, the IMA was ligated 1 cm from the aorta to avoid damaging the nerves.
  Arms: not preserving the left colic artery

SUMMARY:
To evaluate the influence to the blood supply of the anastomosis and the harvest of the No. 253 lymph nodes in different surgical methods--- preserving the left colic artery (LCA) and resect the No. 253 lymph node specifically in the radical resection of rectal carcinoma or dividing at the root of the inferior mesenteric artery (IMA) in the radical resection of rectal carcinoma.

DETAILED DESCRIPTION:
Methods: The patients who got rectal carcinoma are divided into two groups. Both groups will receive the radical resection of rectal carcinoma. We preserve the left colic artery and resect the No. 253 lymph node specifically in Group A and divide at the root of the inferior mesenteric artery in Group B, We insert a trocar into the arterial arcade at the proximal site of the anastomosis and measure the blood pressure of the arterial arcade in the operation, which can reflect the blood supply of the anastomosis. Besides, We will measure the length of the colon from the anastomosis to the level of the root of the IMA. Expecting Results：The blood pressure of the arterial arcade in Group A will be higher than that in Group B. And the patients in Group A will have less chance to get anastomotic fistula. Expecting Conclusions: Preserving the LCA and resecting the No. 253 lymph node specifically in the radical resection of rectal carcinoma can improve the blood supply of the anastomosis and decrease the incidence of anastomotic fistula, and won't affect the harvest of the No. 253 lymph node.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming to FirstJilinU diagnosed rectum cancer by endoscopy and pathology.
* The rectum cancer is the first malignant neoplasm the patient has got.
* The cancer is solitary, and is 3cm to 20cm to the anus.
* The surgical method is limited to Dixon.

Exclusion Criteria:

* Being in the acute phase of inflammation before operation and emergency surgery.
* Patients receiving steroid medication or preoperative radiotherapy。
* Discovering macrometastasis before or in the operation.
* The rectum cancer that can't be radical resected.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2013-02; Primary Completion 2014-09 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Suo, Dr., Study Chair — Department of Gastrointestinal Surgery, First Hospital of Jilin University, Changchun, China.
Locations (1):
- First Hospital of Jilin University, Changchun, Jilin, China

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 69 Chinese patients from the First Hospital of Jilin University were recruited for the study between February 2013 and December 2013 .
Pre-assignment Details: 69 patients initially considered for the study, 11 were excluded because they didn't meet the including criteria. The remaining 58 patients were informed with regard to the study, but they remained blinded to the type of operative technique they would receive. Ultimately, one patient declined to participate in the study.
Groups:
- High Ligation of IMA: We performed the high ligation of the inferior mesenteric artery during the rectal surgery.
  not preserving the left colic artery: The root of the IMA was exposed and the fatty tissue around the root of the IMA was swept in order to maximize the lymph node retrieval rate. Subsequently, the IMA was ligated 1 cm from the aorta to avoid damaging the nerves.
- Left Colic Artery Preserved: We preserve the left colic artery and resect the No. 253 lymph node during the rectal surgery.
  preserving the left colic artery: The root of the inferior mesenteric artery(IMA) was carefully dissected and the artery wall was exposed all the way to the bifurcation of the left colic artery(LCA) and the superior rectal artery (SRA), exposing the LCA from its root until the inferior mesenteric vein (IMV) was recognized. Subsequently, dissection was continued along the IMV up to the level of the root of the IMA. Then the sigmoid mesentery was transected from the root of the IMA to the IMV, and the IMV and the root of the SRA were ligated. Finally, the adipose tissue with the lymph nodes in the area surrounded by the IMA, IMV, and LCA was dissected, with preservation of the LCA .
Period: Overall Study
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved
Started | 29 | 28
Completed | 29 | 28
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved | Total
Number analyzed (Participants) | 29 | 28 | 57
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 17 | 39
  >=65 years | 7 | 11 | 18
Age, Continuous [Mean (Full Range); unit: years] | 59.3 [34 to 71] | 62.1 [45 to 81] | 60.7 [34 to 81]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 24
  Male | 16 | 17 | 33
Region of Enrollment [Number; unit: participants]
  China | 29 | 28 | 57

OUTCOME MEASURES:

1. Primary Outcome: The Blood Pressure of the Arterial Arcade
Time Frame: after ligating the inferior mesentric artery or superior rectal artery
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved
Number analyzed (Participants) | 29 | 28
mmHg | 42.31 (1.85) | 48.50 (2.48)

2. Secondary Outcome: Distal Colon Length
Time Frame: after digestive tract reconstruction
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved
Number analyzed (Participants) | 29 | 28
cm | 20.03 (3.27) | 21.29 (4.91)

3. Other Pre Specified Outcome: Systemic Blood Pressure
Time Frame: after ligating the inferior mesentric artery and measuring the blood pressure of the marginal artery of distal colon
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved
Number analyzed (Participants) | 29 | 28
mmHg | 82.86 (10.17) | 81.21 (11.58)

ADVERSE EVENTS:
Arm/Group | High Ligation of IMA | Left Colic Artery Preserved
Serious Adverse Events (participants affected / at risk) | 3/29 | 1/28
Other Adverse Events (participants affected / at risk) | 0/29 | 0/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | High Ligation of IMA (N=29) | Left Colic Artery Preserved (N=28)
anastomotic leakage (Surgical and medical procedures) | 3 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes